CLINICAL TRIAL: NCT00468624
Title: A Study of the Relationship Between Serum Growth Hormone (GH) and Insulin-Like Growth Factor One (IGF-I) in Patients With Severe Adult Growth Hormone Deficiency (AGHD)
Brief Title: Effect of Pegvisomant on GH/IGF-I Relationship in GHD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment completed
Sponsor: The Christie NHS Foundation Trust (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 04_ENDO_41
Record Dates: First submitted 2007-05-02; First posted 2007-05-03 (Estimated); Last update posted 2007-05-03 (Estimated); Status verified 2007-05

CONDITIONS: Severe Adult Growth Hormone Deficiency
Keywords: Growth hormone; insulin-like growth factor 1; pegvisomant
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — pegvisomant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: pegvisomant/placebo loading dose 80mg sc, thereafter 20mg daily for 2 weeks
Procedure: GH sampling - every 20 min over 24 hours after each limb (pegvisomant/placebo)
Procedure: blood sampling before and after pegvisomant/placebo
Procedure: arginine stimulation test after each limb

SUMMARY:
Approximately 50% of middle-aged patients with severe AGHD have a normal age-related serum IGF-I. It remains unclear if in these individuals serum IGF-I is GH dependent or independent. This study compared the relationship between GH and serum IGF-I in two cohorts of male patients with severe AGHD; one with normal and the other with subnormal age-related serum IGF-I values. The GH receptor antagonist - pegvisomant was be used to specifically inhibit GH action and the changes in markers of the GH axis, such as serum IGF-I, IGFBP-3, GH and GHBP were measured.

DETAILED DESCRIPTION:
There is an increasing reliance on serum insulin-like factor-I (IGF-I) in the management of disturbances of the growth hormone (GH) axis. IGF-I is predominantly, but not exclusively, regulated by GH secreted from the pituitary, with the majority of circulating IGF-I being hepatic in origin.

In parallel with the age-related decline in GH secretion, circulating levels of IGF-I fall with age (1). For a given GH level women have lower serum IGF-I levels than men, indicative of a relative GH resistance (1,2). Nutrition-related factors are known to affect GH, IGF-I and their relationship. Obesity is associated with low GH production, but increased GH sensitivity resulting in relatively high IGF-I for given GH (3-6). Deprivation of important nutrients during fasting is known to stimulate GH, whilst reducing IGF-I (7-9). In vitro studies demonstrated complex role of insulin in IGF-I generation. Insulin stimulates hepatic IGF-I production directly by increasing IGF-I mRNA synthesis and indirectly by enhancing the effect of GH (10,11). By decreasing insulin-like growth factor 1 and 2 (IGFBP1-2), insulin may also affect bioavailability of IGF-I (12-13).

In acromegaly, IGF-I is an important marker for diagnosis and monitoring of disease activity. If patients are treated with a GH receptor antagonist, IGF-I becomes the only useful biochemical marker for monitoring disease activity.

GH deficiency in adults is associated with increased morbidity (14-16). In patients with pituitary disease there has been great progress in the recognition and treatment of this disorder. There is increasing awareness of GH deficiency, not only as a complication of the long-recognised causes of hypopituitarism, but also in the setting of traumatic brain injury and subarachnoid haemorrhage (17). The phenotype of severe adult GHD has been described but many of the features lack specificity and biochemical confirmation of the diagnosis is necessary. The Port Stevens consensus on severe adult GHD relies on the measurement of stimulated GH secretion for confirmation of the diagnosis with a peak GH of <3 µg/L, in one or two stimulation tests, depending on the number of other pituitary hormone deficiencies (18) GH replacement therapy relies on measurement of serum IGF-I for dose titration, with the biochemical goal being of placing circulating IGF-I within age- and gender-related reference range, preferably between 0 and +1 SDS (19). The Port Stephens consensus recognises the apparent paradox that approximately 50% of middle-aged patients diagnosed with severe GHD by a peak stimulated GH levels of <3 µg/L have a pre-treatment IGF-I within the reference range. In untreated severe GHD of adult onset and predominately in men, serum IGF-I may even be in the upper half of reference range. In other words, before treatment these patients already have an IGF-I that would be regarded as satisfactory response to GH replacement therapy. Prima facia, it is difficult to reconcile a serum IGF-I within the reference range and a diagnosis of GHD. Inevitably, it poses the question if factors other than GH are regulating circulating IGF-I levels in such patients.

Pegvisomant is a GH analogue that binds to, but does not activate the GH receptor and has been shown to normalise IGF-I in up to 97% of patients with acromegaly (20). We used pegvisomant to study the relationship between GH and IGF-I in patients with severe adult GHD and investigate whether IGF-I in such patients, is particularly GH-dependent.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Confirmed severe AGHD
* GH response <9 mU/l (preferably <4) to insulin-induced hypoglycaemia or glucagon stimulation test plus (These tests will have taken place as part of routine management).
* Full, stable pituitary replacement therapy
* Willing to provide informed consent

Exclusion Criteria:

* Unwilling to provide written consent
* Current GH therapy
* Pharmacological doses of glucocorticoids
* Any acute illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2004-12; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
change in IGF-I | 2 weeks per limb

SECONDARY OUTCOMES:
change in basal and stimulated GH Change in IGFBP-3 Change in GHBP | 2 weeks per limb

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Trainer, MD FRCP, Principal Investigator — Christie Hospital NHS
Locations (1):
- Christie Hospital NHS Trust, Manchester, United Kingdom

REFERENCES:
- [Background] 1. Svensson J, Johannsson G, Bengtsson BA 1997 Insulin-like growth factor-I in growth hormone-deficient adults: relationship to population-based normal values, body composition and insulin tolerance test. Clin Endocrinol (Oxf) 46:579-586 2. Veldhuis JD 1996 Gender differences in secretory activity of the human somatotropic (growth hormone) axis. Eur J Endocrinol 134:287-295 3. Caufriez A, Golstein J, Lebrun P, Herchuelz A, Furlanetto R, Copinschi G 1984 Relations between immunoreactive somatomedin C, insulin and T3 patterns during fasting in obese subjects. Clin Endocrinol (Oxf) 20:65-70 4. Copeland KC, Colletti RB, Devlin JT, McAuliffe TL 1990 The relationship between insulin-like growth factor-I, adiposity, and aging. Metabolism 39: 584-587 5. Yamamoto H, Kato Y 1993 Relationship between plasma insulin-like growth factor I (IGF-I) levels and body mass index (BMI) in adults. Endocr J 40:41-45 6. Rasmussen MH, Ho KK, Kjems L, Hilsted J 1996 Serum growth hormone-binding protein in obesity: effect of a short-term, very low calorie diet and diet-induced weight loss. J Clin Endocrinol Metab 81:1519-1524 7. Ho KY, Veldhuis JD, Johnson ML, Furlanetto R, Evans WS, Alberti KG, Thorner MO 1988 Fasting enhances growth hormone secretion and amplifies the complex rhythms of growth hormone secretion in man. J Clin Invest 81:968-975 8. Maccario M, Aimaretti G, Grottoli S, Gauna C, Tassone F, Corneli G, Rossetto R, Wu Z, Strasburger CJ, Ghigo E 2001 Effects of 36 hour fasting on GH/IGF-I axis and metabolic parameters in patients with simple obesity. Comparison with normal subjects and hypopituitary patients with severe GH deficiency. Int J Obes Relat Metab Disord 25:1233-1239 9. Darzy KH, Murray RD, Gleeson HK, Pezzoli SS, Thorner MO, Shalet SM 2006: The impact of short-term fasting on the dynamics of 24-hour growth hormone (GH) secretion in patients with severe radiation-induced GH deficiency.J Clin Endocrinol Metab. 91(3):987-94. 10. Boni Schnetzler M, Schmid C, Meier PJ, Froesch ER 1991 Insulin regulates insulin-like growth factor I mRNA in rat hepatocytes, Am J Physiol 260: 846-51. 11. Leung KC, Doyle N, Ballesteros M, Waters MJ, Ho KK. 2000 Insulin regulation of human hepatic growth hormone receptors: divergent effects on biosynthesis and surface translocation, J Clin Endocrinol Metab 85:4712-20. 12. Cox GN, McDermott MJ, Merkel E, Stroh CA, Ko SC, Squires CH, Gleason TM, Russell D. 1994 Recombinant human insulin-like growth factor (IGF)-binding protein-1 inhibits somatic growth stimulated by IGF-I and growth hormone in hypophysectomized rats, Endocrinology 135: 1913-20. 13. Wolf E, Lahm H, Wu M, Wanke R,. Hoeflich A, 2000 Effects of IGFBP-2 overexpression in vitro and in vivo, Pediatr Nephrol 14: 572-8. 14. Bates JA, Van't Hoff W, Jones PJ, Clayton RN. 1996 The effect of hypopituitarism on life expectancy. J Clin Endocrinol Metab 81:1169-72 15. Rosen T, Bengtsson B-A. 1990 Premaature mortality due to cardiovascular disease in hypopituitarism. Lancet 336: 285-8 16. Tomlinson JW, Holden N, Hills RK, Wheatley K, Clayton RN, Bates AS, Sheppard MC, Stewart PM. Association between premature mortality and hypopituitarism. West midlands prospective hypopituitary study group. 2001 Lancet 357:425-31. 17. Aimaretti G, Ambrosio MR, Di Somma C, Fusco A, Cannavo S, Gasperi M, Scaroni C, De Marinis L, Benvanga S, degli Uberti EC, Lombardi G, Mantero F, Martino E, Giordano G, Ghigo E. Traumatic brain injury and subarachnoid haemorrhage are conditions at high risk for hypopituitarism: screening study at 3 months after the brain injury. 2004 Clin Endo (Oxf.) 61(3):320-6 18. Consensus Guidelines for the Diagnosis and Treatment of Adults with Growth Hormone Deficiency: Summary Statement of the Growth Hormone Research Society Workshop on Adult Growth Hormone Deficiency 1998 JCE&M; 83(2):379-81 19. Mukherjee A, Monson JP, Jonsson PJ, Trainer PJ, Shalet SM 2003 Seeking the optimal target range for insulin-like growth factor I during the treatment of adult growth hormone disorders. J Clin Endocrinol Metab 88:5865-5870 20. Van der Lely AJ, Hutson RK, Trainer PJ, Besser GM, Barkan AL, Katznelson L, Klibanski A, Herman-Bonert V, Melmed S, Vance ML, Freda PU, Stewart PM, Friend KE, Clemmons DR, Johannsson G, Stavrou S, Cook DM, Phillips LS, Strasburger CJ, Hackett S, Zib KA, Davis RJ, Scarlett JA, Thorner MO. 2001 Long-term treatment of acromegaly with pegvisomant, a growth hormone receptor antagonist. Lancet 358: 1754-59